CLINICAL TRIAL: NCT03176056
Title: Low Carbohydrate Diet for Type 2 Diabetes Mellitus
Brief Title: The Effectiveness of Low Carbohydrate Diet in Reducing Polypharmacy for Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201504032RINA
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Low carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet (Experimental): Low carbohydrate diet limits carbohydrate <=90g/day
  Interventions: Dietary Supplement: Low carbohydrate diet
- Calori restricted diet (Active Comparator): Traditional diabetic diet
  Interventions: Dietary Supplement: Calori restricted diet

INTERVENTIONS:
Dietary Supplement: Low carbohydrate diet — For the LCD group, the daily carbohydrate intake was limited to less than 90g, without any restriction to total energy. The concept of a LCD was introduced and an educational 15 g equivalent carbohydrate food list was provided. The easy conversion method is that 15 g equivalent carbohydrate =1/4 bowel of rice= 1/2 bowel of noodle = 1 slice of toast = 3 soup-spoon of oats = one bowl of fruit =1/2 regular size banana= one glass of milk = 3 dumplings. Less than two equivalent 15g-carbohydrate intakes per meal were advised.
  Arms: Low carbohydrate diet
Dietary Supplement: Calori restricted diet — For the calori restricted diet group, the target total calorie intake was calculated by multiplying the ideal body weight by 25 kcal/kg for those with a BMI in the range 18.5 to 24, 20 kcal/kg for obese subjects with a BMI > 24 and 30 kcal/day for underweight subjects with a BMI <18.5. The macronutrient percentage was 50-60% for carbohydrate, 1.0-1.2 g/kg for protein and fat ≦30%.
  Arms: Calori restricted diet

SUMMARY:
This study determines whether an educational intervention with a 90 g/day LCD is safe, effective and has good compliance for poorly controlled type 2 diabetes patients.

DETAILED DESCRIPTION:
Poorly controlled type 2 diabetic men and women, aged between 20 and 80 years, with HbA1c≧ 7.5% (58mmol/mol) in the previous 3 months participated in this randomized controlled 18-month trial at a medical center. Patients were randomly assigned to the interventional group and given a 90g/day low carbohydrate diet (LCD) or the controlled group, which maintained a standard calorie-restricted diet (CRD). All patients received periodic educational intervention and were monitored for weight, body composition, waist girth, hip girth, thigh girth, pre- and post-prandial serum glucose, HbA1c, lipid profile(Cholesterol, Triglyceride. HDL, LDL, sdLDL), renal function, microalbumin/cre, carotid intima-media thickness (IMT),and medication effect score (MES).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosis ≧ 1 year
* poorly controlled with HbA1c≧ 7.5% in the previous 3 months.
* aged 20 to 80
* without or with treatment [ oral hypoglycemic agents (OHA) and/or insulin treatment)

Exclusion Criteria:

* pregnancy or lactating women
* impaired renal function with serum creatinine ≧ 1.5 mg/dl
* abnormal liver function [alanine aminotransferase (ALT), aspartate aminotransferase (AST), ≧ 3 times the normal upper limit) or liver cirrhosis
* significant heart diseases (unstable angina, unstable heart failure)
* frequent gout attacks (≧ 3 times/year)
* participation in other weight loss programs or the use of weight-reducing drugs
* eating disorders
* could not complete the questionnaire
* poor compliance to protocol.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
The improvement of glycemic control status | measured at baseline and every 3 months for 18 months after intervention
  The reduction of HbA1c, fasting and 2-h glucose over the 18 months after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.
The reduction of medication effect score (MES) | measured at baseline and every 3 months for 18 months after intervention
  The MES assessed the overall utilization of hypoglycemic agents. The percentage of the maximum daily dose for each medication was multiplied by an adjustment factor and these products were summed to produce the final MES value. A higher MES value denoted a greater use of medication. The minimum score is 0 and without maximum score.The lower, the better. The reduction of MES over the 18 months after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.

SECONDARY OUTCOMES:
The improvement of lipid profile | measured at baseline and every 3 months for 18 months after intervention
  The reduction of total cholesterol, triglyceride, LDL and the increment of HDL after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.
The improvement of small dense low density lipoprotein (sdLDL) | measured at baseline and every 6 months for 18 months after intervention
  The reduction of sdLDL after intervention.The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.
The maintenance of renal function | measured at baseline and every 3 months for 18 months after intervention
  The change of serum creatinine after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.
The improvement of microalbuminuria. | measured at baseline and 18 month after intervention
  The reduction of microalbumin/creatine ratio after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.
The improvement of carotid intima-media thickness (IMT) | measured at baseline and 18 month after intervention
  The reduction of carotid IMT after intervention. The analysis of generalized estimating equation parameters and empirical standard error estimates for the time-group difference over 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Ying Chen, MD, MHSc, Study Chair — National Taiwan University Hospital and National Taiwan University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-07-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT03176056/Prot_000.pdf